CLINICAL TRIAL: NCT03914040
Title: Interprofessional Learning and Simulation Versus Traditional Course on Healthy Aging: a Randomized Control Trial
Brief Title: Effectiveness of Interprofessional Learning and Simulation on Healthy Aging in Undergraduate Medical and Nursing Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Massimiliano Panella, Department of traslational medicine, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IPSE_UPO students
Record Dates: First submitted 2019-04-01; First posted 2019-04-12 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Healthy Aging; Interprofessional Relations; Education, Professional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPSE program (Experimental): IPSE is conceptually divided in two phases: 1) pre-immersion preparation, 2) immersion.
  Interventions: Other: IPSE program
- Traditional course (No Intervention): Participants in the control group will receive the current face-to-face course.

INTERVENTIONS:
Other: IPSE program — 1. Pre-immersion preparation. A self-study course will be offered about lifestyle modification. Some readings will be suggested to introduce students to the concepts of health promotion and prevention of metabolic syndrome.
  2. Immersion. Four different learning methods will be provided: I) four hours of didactic lectures followed by group discussion, II) four hours per student of role playing, III) 30' per students of standardized patient experiences and IV) 30' per students of a new immersive advanced simulation learning environment (e-REAL). Four case-studies will be used to create scenarious, including woman with menopause weight gain, obese young adult, obese child and adult with unhealthy behaviours.
  Arms: IPSE program

SUMMARY:
Aging population is an important public health issue and require coordinated and comprehensive response. Medical and nursing schools need to address challenges in health care delivery, and interprofessional simulation-based education (IPSE) provides realistic learning experiences in which interprofessional communication, roles and teamwork can be developed and assessed.

The study aims to examine the effectiveness of delivering an IPSE program versus traditional course to nursing and medical students. The primary outcome is improved communication skills, assessed by Communication Skill Attitude Scale (CSAS) divided in two subscales: Positive Attitude Scale (PAS) and Negative Attitude Scale (NAS).

DETAILED DESCRIPTION:
Design: this is a randomized, controlled study. Eligible participants will be randomly allocated to intervention group (IPSE) or control group (traditional course) in a 1:1 ratio. The investigator will use a block size of four with no stratification: for each block of 4 students, a different random ordering of 2 assignments to each treatment will be produced. A table of random numbers will be used to produce 2 randomization lists: one for nursing students and one for medical students.

Setting and participants: the study will be performed at the Università del Piemonte Orientale (Italy). In this study, second-year student volunteers from the Nursing School and fourth and fifth-year student volunteers from the School of Medicine will be recruited through an information session.

Intervention: IPSE program is divided in two phases: 1) a self-study course will be offered about lifestyle modification, 2) four different learning methods: didactic lecture, role playing, standardized patient and a new immersive advanced simulation learning environment will be provided.

Data collection: demographic data (gender, age, education) will be gathered to obtain a basic profile of participants prior to allocation. Before the randomization and after the completion of the program, each participant will complete the evaluation session.

Sample size calculation: a minimal total study sample size of 60 (24 nursing and 36 medical students) would be required to provide 80% power to reject the null hypothesis that no difference existed between the two research arms in NAS/PAS score, with a two-sided type 1 error of 5%. To balance the sample size of the two groups, the investigator decided to recruit the same number of nursing and medical students: 36 participants for each group. With a 10% allowance for students lost at follow up, a sample size of 80 students would be required and will be used.

Analyses: all analyses will be based on the Intention-To-Treat (ITT) approach. Students who do not start intervention or only complete the 25% of the course will not be included in the analysis. Descriptive statistical analyses will be conducted separately for each student group using the information collected at baseline. For categorical variables, number and percentage of participants in each category will be reported while, for normally distributed continuous variables, the mean and Standard Deviation values will be calculated. If the data are not normal, the investigator will use median and interquartile range. Subsequently, the analyses will be conducted categorizing the continuous variables and joining levels of ordinal variables to avoid the occurrence of scattered data phenomena.

In order to evaluate baseline differences between nursing and medical students, approximate (Chi square) or exact (Fisher) association tests will be performed for categorical variables while, for numeric ones, the investigator will use the independent T-test(parametric) or the Mann-Whitney U test (nonparametric). The obtained p value values will be reported.

The individual response profiles of primary outcomes will be implemented. Then, subjects will be categorized into two groups: successful if they increase positive scores/decrease negative scores and unsuccessful if they decrease positive scores/increase negative scores. The association with these binary outcomes and the recorded variables will be evaluated with appropriate tests (Chi-square, Fisher Exact, T, Mann-Withey). For each outcome the Relative Risks will be calculated with the respective 95% Confidence Interval using a Poisson regression with a robust error variance.

Study data will gather and manage with REDCap31 electronic data-capture tools, and the analyses will be performed by using SAS version 9.4.

ELIGIBILITY:
Inclusion Criteria:

* second-year nursing students,
* fourth and fifth-year medical students.

Exclusion Criteria:

* students who had already failed the course in a previous year.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Communication skills. | From baseline to one month.
  Communication Skill Attitude Scale (CSAS).CSAS is a 26-item questionnaire in two dimensions that has been developed to measure positive and negative attitudes towards learning communication skills. Each of the two subscales consists of 13 items, the Positive Attitude Scale (PAS) and the Negative Attitude Scale (NAS).

SECONDARY OUTCOMES:
Students' perception of the professional role of physician and nurse. | From baseline to one month
  The measurement tool is the semantic differential test. It consists of a series of 16 bipolar adjective-pair scales for measuring psychological meanings related to three concepts: "me as a medical or nursing student", "physician using lifestyle medicine approach" and "nurse using lifestyle medicine approach".The meaning of the concept is measured by individual, selecting a point along a seven-point scale. The point selected indicates both the quality and intensity of the participant's subjective assessment of the association between the adjective pair and the related concept.

OTHER OUTCOMES:
Students' self-confidence about learning in simulation. | up to 1 week after intervention
  The Student Satisfaction and Self-Confidence in Learning Scale (SCLS). A total of 13 items assess the attitudes toward satisfaction with instruction and self-confidence in learning in simulation. For each item, participants indicated their personal feelings about a statement that described their own attitudes or beliefs. Response options are 1) strongly disagree, 2) disagree, 3) undecided, 4) agree, and 5) strongly agree using a Likert-style scale. Scores are calculated by summing responses; higher scores indicate more satisfaction and more self-confidence, respectively.
Students' perception about learning in simulation | up to 1 week after intervention
  Simulation Design Scale (SDS). A total of 20 items assess perceptions of objectives, information, support, problem solving, feedback, and fidelity in simulation. For each item, participants indicate their perceptions about a statement that described the presence of simulation design features. Response options for statements related to presence of simulation design features are 1) strongly disagree, 2) disagree, 3) undecided, 4) agree, 5) strongly agree, and NA) not applicable using a Likert-style scale. Scores are calculated by summing responses; higher scores represent increased recognition of design features in simulation.
Students' perception of the presence of educational best practices in simulation | up to 1 week after intervention
  Educational Practices Questionnaire (EPQ).The instrument consists in 16 items. For each item, participants indicated their perceptions about a statement that described presence of educational best practices. Items are rated on a Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree). Scores are calculated by summing responses; higher scores represent increased recognition of educational best practices in simulation.

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Panella, Principal Investigator — Dipartimento di medicina traslazionale-Università degli studi del piemonte orientale
Locations (1):
- Università del Piemonte Orientale, Novara, Italy

IPD SHARING:
Plan to Share IPD: No
Study protocol and final report will be submitted to peer-reviewed journal for possible publication.